CLINICAL TRIAL: NCT01928875
Title: Comparison of Adequacy of Anesthesia Monitoring With Standard Clinical Practice During Routine General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 123.04-2012-GES-0009
Record Dates: First submitted 2013-08-19; First posted 2013-08-27 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Surgical Procedure, Unspecified

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adequacy of Anesthesia (AoA) Monitoring (Experimental): Adequacy of Anesthesia monitoring with SPI and Entropy
  Interventions: Device: AoA Monitoring
- Routine (Standard) Anesthesia Monitoring (Active Comparator)
  Interventions: Device: Routine (Standard) Anesthesia Monitoring

INTERVENTIONS:
Device: AoA Monitoring — Monitoring with Entropy and SPI parameters during surgery
  Arms: Adequacy of Anesthesia (AoA) Monitoring
Device: Routine (Standard) Anesthesia Monitoring — Standard of care monitoring
  Arms: Routine (Standard) Anesthesia Monitoring

SUMMARY:
The purpose of this study is to demonstrate that using Surgical Pleth Index (SPI) and Entropy in adjunct to other clinical information decreases the occurrence rate of inadequate anesthesia events, bradycardia and hypotension in comparison to standard clinical practice during anesthesia. Adequacy of Anesthesia (AoA) monitoring comprises the use of both Entropy and SPI measurements. Adequacy of anesthesia will be monitored using non-invasive blood pressure, blood oxygen saturation (SpO2), ECG, and neuromuscular transmission (NMT).

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Age 18-80 years of age
* Surgery that is expected to last at least 2 hours under general anesthesia with endotracheal tube

Exclusion Criteria:

* Any subject that meets the definition of vulnerable subject as defined in ISO 14155:2011
* Per ISO 14155:2011, a vulnerable subject is defined as an individual whose willingness to volunteer in a clinical investigation could be unduly influenced by the expectation, whether justified or not, of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate
* Any subject with a cardiac pacemaker
* Any subject with atrial fibrillation at the time of obtaining the baseline values
* Any subject with more than 5 ventricular extra systoles/minute at the time of obtaining the baseline values
* Any subject who needs invasive blood pressure measurement
* Any subject who show hemodynamics that would have qualified for being considered as a sign of inadequate anesthesia already at baseline:
* Mean blood pressure below 60 mmHg or above 100 mmHg
* HR below 45 /min or above 100/min
* Any subject with epidural anesthesia or analgesia during the surgery. Epidural catheter may be placed pre-operatively, and used in the PACU, but not during the surgery
* Any subject having surgery that requires prone position
* Any subject with very high body mass index (>35) because of incompatibility with the target controlled anesthesia models used
* Any subject with known allergies to the specific anesthetic agents/ analgesic drugs intended for use in their surgeries
* Any subject with laryngeal mask airway
* Any subject who requires neuromuscular blocking agent infusion
* Any subject who is going to have major surgery with a high risk of extensive blood loss
* Any subject with known chronic use of opioids

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2013-12; Primary Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of hemodynamic instability | Participants will be followed for the duration of their surgery
  Incidence of hemodynamic instability including hypertension, hypotension, tachycardia, and bradycardia

CONTACTS AND LOCATIONS:
Locations (4):
- Tampere University Hospital, Tampere, Finland
- University Hospital Schleswig-Holstein, Kiel, Germany
- University of Szeged, Szeged, Hungary
- University of Amsterdam, Amsterdam, Netherlands

REFERENCES:
- [Derived] Gruenewald M, Harju J, Preckel B, Molnar Z, Yli-Hankala A, Rosskopf F, Koers L, Orban A, Bein B; AoA Study Group. Comparison of adequacy of anaesthesia monitoring with standard clinical practice monitoring during routine general anaesthesia: An international, multicentre, single-blinded randomised controlled trial. Eur J Anaesthesiol. 2021 Jan;38(1):73-81. doi: 10.1097/EJA.0000000000001357. PMID 33074943